CLINICAL TRIAL: NCT05335369
Title: A Pilot Randomized Controlled Trial of a Patient-centered Communication Tool (UR-GOAL) for Older Patients With Acute Myeloid Leukemia, Their Caregivers, and Their Oncologists
Brief Title: A Patient-Centered Communication Tool (UR-GOAL) Versus Usual Care for Older Patients With Acute Myeloid Leukemia, Their Caregivers, and Their Oncologists
Acronym: UR-GOAL 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Kah Poh Loh, Associate Professor - Department of Medicine, Hematology/Oncology (SMD), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UOCPC22010
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; communication; shared decision making; older adults; geriatric hematology
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Communication

STUDY DESIGN:
Intervention Model Description: The UR-GOAL 1) conducts assessments of fitness, 2) elicits patient values via Best-Worst Scaling, and 3) elicits preferences for prognostic information and assesses prognostic awareness. The tool also includes an AML educational video.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Usual care
- UR-GOAL (Experimental): UR-GOAL helps conducts assessments of fitness, elicits patient values via Best-Worst Scaling, and elicits preferences for prognostic information and assesses prognostic awareness. The tool also includes an AML educational video.
  Interventions: Behavioral: UR-GOAL

INTERVENTIONS:
Behavioral: UR-GOAL — UR-GOAL helps conducts assessments of fitness, elicits patient values via Best-Worst Scaling, and elicits preferences for prognostic information and assesses prognostic awareness. The tool also includes an AML educational video.
  Arms: UR-GOAL

SUMMARY:
The objective of this study is to conduct a pilot randomized trial to evaluate the preliminary efficacy of the UR-GOAL tool in improving SDM and communication between 100 older patients with AML and their oncologists.

DETAILED DESCRIPTION:
The investigators have developed a patient-centered communication tool (University of Rochester-Geriatric Oncology assessment for Acute myeloid Leukemia or UR-GOAL) that 1) conducts assessments of fitness, 2) elicits patient values via Best-Worst Scaling, and 3) elicits preferences for prognostic information and assesses prognostic awareness. The tool also includes an AML educational video. The investigators have refined the tool based on feedback from stakeholders consisting of older patients with cancer, caregivers, and oncologists. This was further adapted in a qualitative study of 15 older patients with AML. In a single arm pilot study, the investigators have demonstrated feasibility of recruiting older patients with newly diagnosed AML to a single arm study, as well as their caregivers and oncologists.

ELIGIBILITY:
Inclusion Criteria:

Patients

1. Age ≥60 years
2. Newly diagnosed AML or being worked up for possible AML
3. Able to provide informed consent
4. Agreement of their oncologist to participate in the study
5. English-speaking

If patients screen positive for cognitive impairment on the Mini-Cog test performed as part of the baseline assessment, they can still enroll if they are able to provide informed consent and have decision making capacity as determined by their treating oncologist

Caregivers

1. Selected by the patient when asked if there is a "family member, partner, friend or caregiver [age 21 or older] with whom the patient discuss or who can be helpful in health-related matters;" patients who cannot identify such a person ("caregiver") can be eligible for the study. A caregiver need not be someone who lives with the patient or provides direct hands-on care. A caregiver can be any person who provides support (in any way) to the patient
2. Able to provide informed consent
3. English-speaking

Oncologists

1. A practicing oncologist
2. At least one of their patients are recruited to the study
3. English-speaking

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Shared Decision Making | Within 1-4 weeks after treatment initiation
  A 9-item reliable questionnaire assessing patient satisfaction with the medical decision-making process, range 0-45, higher score indicates greater shared decision making

SECONDARY OUTCOMES:
Patient-Centered Communication in Cancer Care (PCC-Ca-36) | Within 1-4 weeks after treatment initiation
  A 36-item questionnaire assessing patient-centered communication in six domains: exchanging information, making decisions, fostering healing relationships, enabling patient self-management, managing uncertainty, and responding to emotions. Scores in each domain range from 1-5, higher scores indicate better communication. Scores are reported in each domain and overall.

CONTACTS AND LOCATIONS:
Overall Officials: Kah Poh Loh, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other investigators if requested. The investigators will publish our study protocol. Published papers will be made available in portable document format.
Supporting Information: Study Protocol
Time Frame: The data will be available for 7 years after study completion

REFERENCES:
- [Background] DuMontier C, Loh KP, Soto-Perez-de-Celis E, Dale W. Decision Making in Older Adults With Cancer. J Clin Oncol. 2021 Jul 1;39(19):2164-2174. doi: 10.1200/JCO.21.00165. Epub 2021 May 27. No abstract available. PMID 34043434
- [Background] Loh KP, Abdallah M, Kadambi S, Wells M, Kumar AJ, Mendler JH, Liesveld JL, Wittink M, O'Dwyer K, Becker MW, McHugh C, Stock W, Majhail NS, Wildes TM, Duberstein P, Mohile SG, Klepin HD. Treatment decision-making in acute myeloid leukemia: a qualitative study of older adults and community oncologists. Leuk Lymphoma. 2021 Feb;62(2):387-398. doi: 10.1080/10428194.2020.1832662. Epub 2020 Oct 11. PMID 33040623
- [Derived] Jensen-Battaglia M, LoCastro M, Oh H, Sanapala C, Flannery M, Mendler JH, Liesveld J, Huselton E, Loh KP. Patient-oncologist discussion of treatment decisions: Exploring the role of a patient-centered communication tool for older adults with acute myeloid leukemia and their caregivers. J Geriatr Oncol. 2024 Jun;15(5):101716. doi: 10.1016/j.jgo.2024.101716. Epub 2024 Feb 9. No abstract available. PMID 38336521